CLINICAL TRIAL: NCT07145372
Title: A Comparative Study of Diaphragm Relaxation Techniques, Diaphragmatic Breathing Exercises, and Manual Therapy on Pain and Quality of Life in Individuals With Migraine
Brief Title: Diaphragm Relaxation Techniques, Diaphragmatic Breathing Exercises for Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seda Saka (Other)
Responsible Party: Sponsor-Investigator, Seda Saka, Physiotherapist, PhD, Halic University
Organization: Halic University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EH250
Record Dates: First submitted 2025-08-13; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Migraine; Migraine Disease; Manuel Therapy; Diaphragm Relaxation
Keywords: Diaphragm Relaxation; Manual Therapy; Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual therapy group (Experimental): It includes 10 minutes of massage and myofascial release for the trapezius and neck extensors, 10 repetitions of occiput-atlas (C0-C1) joint mobilization, occiput-atlas joint manipulation, mobilization of each segment from C2 to C7 with 10 repetitions each, C2-C7 manipulation, cervicothoracic junction (C7-T1) manipulation, thoracic region (T2-T6) manipulation, and sacroiliac joint manipulation.
  Interventions: Other: Manual therapy
- Diaphragm relaxation group (Experimental): It includes diaphragm manual release techniques and a diaphragmatic breathing exercise program
  Interventions: Other: Diaphragmatic relaxation technique
- Control group (Sham Comparator): This group was given a home exercise program consisting of shoulder girdle range of motion (ROM) exercises that do not affect the cervical region.
  Interventions: Other: Shoulder ROM exercise

INTERVENTIONS:
Other: Manual therapy — It includes 10 minutes of massage and myofascial release for the trapezius and neck extensors, 10 repetitions of occiput-atlas (C0-C1) joint mobilization, occiput-atlas joint manipulation, mobilization of each segment from C2 to C7 with 10 repetitions each, C2-C7 manipulation, cervicothoracic junction (C7-T1) manipulation, thoracic region (T2-T6) manipulation, and sacroiliac joint manipulation.
  Arms: Manual therapy group
Other: Diaphragmatic relaxation technique — It includes diaphragm manual release techniques and a diaphragmatic breathing exercise program
  Arms: Diaphragm relaxation group
Other: Shoulder ROM exercise — This group was given a home exercise program consisting of shoulder girdle range of motion (ROM) exercises that do not affect the cervical region.
  Arms: Control group

SUMMARY:
Migraine is a neurological disease characterized by recurring headaches. It is a significant public health problem of the top reasons for disability throughout the world. This study is planned to compare the effects of relaxation techniques of the diaphragm (midsection), diaphragmatic respiration exercises, and manual therapy applications on the severity and intensity of pain and lquality of life. 42 patients diagnosed with migraine aged between 18 and 60 participated in the study. Patients were divided into 3 groups; diaphragm relaxation group (DG), manual therapy group (MG) and control group (CG). 2 types of evaluation were carried out, one of which was pre-treatment and the other was post-treatment. Visual Analogue Scale (VAS), Megill-Melzack Pain Questionnaire, Headache Impact Test (HITS), and SF-36 Life Quality Scale were used. How long the attacks of patients before and after the treatment lasted and monthly attack numbers were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate voluntarily and having signed informed consent
* Aged between 18 and 60 years
* Diagnosed with migraine
* Not receiving migraine prophylactic treatment
* At least primary school graduate

Exclusion Criteria:

* Using antidepressant medication
* Experiencing other types of headaches alongside migraine
* Undergoing prophylactic treatment for migraine
* Showing signs of vertebral artery or internal carotid artery involvement
* Having vertigo
* Having decompensated blood pressure
* Participated in a neck physiotherapy program within the last 3 months
* Lacking the mental capacity to complete the HIT-6 scale and illiterate
* Pregnant individuals or those who became pregnant during the study period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline and at the end of third week
  A Visual Analog Scale is a simple tool used to measure a person's level of pain or discomfort. It typically consists of a straight line, usually 10 cm long, where one end represents "no pain" and the other end represents "worst imaginable pain." The patient marks a point on the line that reflects their pain intensity.
McGill Pain Questionnaire (MPQ) | Baseline and at the end of third week
  It includes descriptive words categorized into sensory, affective, and evaluative dimensions, allowing patients to provide a comprehensive report of their pain experience. In our study, the score ranges from 0 to 78, with higher scores reflecting greater pain intensity and unpleasantness, meaning worse outcomes.
Headache Impact Test (HIT-6) | Baseline and at the end of third week
  The HIT-6 is a brief questionnaire designed to measure the impact of headaches on a person's daily life. It assesses pain severity, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The scores range from 36 to 78. A higher score indicates a more severe impact of headaches, so higher values reflect worse outcomes.
SF-36 | Baseline and at the end of third week
  It measures overall health-related quality of life. It covers eight domains including physical functioning, bodily pain, general health, vitality, social functioning, emotional role, and mental health. Each domain is scored from 0 to 100, where higher scores represent better health status or quality of life, meaning better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided